CLINICAL TRIAL: NCT01484080
Title: Phase I/II Randomized Clinical Trial of Neoadjuvant Paclitaxel Versus BIBF 1120 Priming Followed by BIBF 1120 Plus Paclitaxel in Early HER-2 Negative Breast Cancer With Proteomic and Dynamic Imaging Correlates
Brief Title: Neoadjuvant Paclitaxel Versus BIBF 1120 Priming Followed by BIBF 1120 Plus Paclitaxel in Early HER-2 Negative Breast Cancer With Proteomic and Dynamic Imaging Correlates
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Collaborators: Hospital Universitario de Fuenlabrada (Other); M.D. Anderson Cancer Center (Other); Hospital Universitari de Bellvitge (Other); Grupo Espanol de Investigacion del Cancer de Mama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNIO-BR-01-2010/GEICAM/2010-10
Record Dates: First submitted 2011-10-21; First posted 2011-12-02 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: BIBF1120+Paclitaxel (Experimental): 2 weeks run-in of BIBF 1120 alone followed by paclitaxel + BIBF 1120 combination
  Interventions: Drug: BIBF + Paclitaxel
- Arm II: Paclitaxel (Active Comparator): Paclitaxel monotherapy treatment will start within 2 weeks after randomization.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: BIBF + Paclitaxel — Priming Period:
  Oral BIBF 1120 will be administered during 2 weeks at the dose determined during the phase-I part that can be combined safely with weekly paclitaxel, on a continuous schedule for 14 days.
  One week washout is planned before starting the treatment phase.
  Treatment Phase:
  Paclitaxel 80 mg/m2 iv on days 1, 8 and 15 + BIBF 1120 recommended dose bid po days 1-21 q 21 days. (BIBF 1120 morning dose is skipped on the paclitaxel administration days).
  Arms: Arm I: BIBF1120+Paclitaxel
Drug: Paclitaxel — Paclitaxel 80 mg/m2 iv on days 1, 8 and 15 q 21 days. A total of 4 cycles will be administered in both arms.
  Arms: Arm II: Paclitaxel

SUMMARY:
The investigators plan to study the efficacy of the combination of weekly paclitaxel + BIBF 1120 in early breast cancer using a neoadjuvant schedule and a randomized phase-II trial design, comparing the efficacy vs. weekly paclitaxel alone, followed by surgery and subsequent standards of care (anthracycline based chemotherapy, radiation or hormonal blockade).

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase I dose-escalation study to assess the safety and tolerability of oral (PO) BIBF 1120 administered with intravenous (IV) paclitaxel (80 mg/m2 on days 1, 8 and 15 every 3 weeks) to patients with breast cancer (see Figure 1 for the study flow chart). BIBF 1120 will be administered twice daily PO for 21 consecutive days (Days 1 to 21) in 3-week cycles (morning dose is skipped on the paclitaxel administration days)

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Patients ≥18 year-old
3. Histological diagnosis of localized breast cancer with primary tumour over 2 cm on its longest diameter (measured by mammography and MRI). Any nodal status is allowed when it is an operable tumour at diagnosis. Multicentricity is allowed.
4. HER 2 negative (Inmunohistochemistry - or + over +++; FISH CISH (-); equivalent to HER2/CEP17 copies under 2: HER2 result ++/+++ needs FISH/CISH confirmation.
5. Measurable disease with a primary lesion >2 cm. by RECIST v1.1 criteria
6. ECOG 0-1
7. Adequate hematologic, renal and hepatic function, defined by the following laboratory results obtained within 14 days prior to randomization/registration:

   * Absolute granulocyte count >1.5 x 109/L
   * Absolute platelet count >100 x 109/L
   * Hemogobin >10 g/dL
   * Serum creatinine >1.5 x UNL or a calculated creatinine clearance >50 ml/min
   * Serum bilirubin <1.25 UNL
   * AST/ALT <1.5 times UL
8. Premenopausal women must be under effective birth control (non-hormone) and continue its use for the duration of the study and even 6 months later.
9. For female with childbearing potential, a negative pregnancy test within the prior 7 days to the study enrolment
10. Life expectancy >6 months

Exclusion Criteria:

1. Metastatic or non-surgical breast cancer (including inflammatory).
2. Locally breast cancer with primary lesion under 2 cm. In case of multicentricity, it will not be admitted in the study unless any lesion would be over this length.
3. Previous or concurrent treatment of any kind for breast cancer: hormonal agents, conventional cytotoxic drugs, radiation therapy, targeted drugs, bisphosphonates, monoclonal antibodies or surgery. Chemoprevention with tamoxifen or raloxifene is allowed as far as the treatment was interrupted upon diagnosis and at least 4 weeks prior to inclusion. Same criteria for post-menopausal hormonal replacement therapy. Hormonal contraceptives should be discontinued.
4. HER-2 positive breast cancer defined as over-expression in Immunochemistry of HER-2 3+ or 2+ with positive FISH/CISH
5. Male patients.
6. Pregnancy, lactation or breastfeeding.
7. Active malignancy at any other side (including contra-lateral synchronous breast cancer) besides non-melanoma skin cancer or ductal/lobular of the breast or cervix in situ carcinoma, colon in situ carcinoma accurately treated as well as any other tumour diagnosis >5 years prior to registration without any sign of progression at present time.
8. Concurrent serious medical conditions such as myocardial infarction within 6 months prior to entry, congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled hypertension (under NYHA criteria), uncontrolled psychotic disorders, serious active infections, active peptic ulcer disease, psychiatric illness, HIV infection, active hepatitis, COPD or any other medical conditions that might be aggravated by treatment or limit compliance.
9. Inability to take oral medication
10. History of malabsorption syndrome
11. Proven allergy to paclitaxel or BIBF 1120.
12. Grade ≥2 peripheral neuropathy.
13. Major surgery within 4 weeks of registration (breast cancer surgery regardless of timing is an exclusion criteria).
14. Inability to comply with the study and follow-up procedures.
15. Anticoagulation therapy (except low-dose heparin and / or wash out with heparin as needed to maintain a permanent intravenous device) or antiplatelet therapy (except for treatment with low doses of aspirin <325 mg per day.
16. History of hemorrhagic or thromboembolic event clinically significant in the last 6 months.
17. Known hereditary predisposition to bleeding or thrombosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response | Within 30 days after surgery
  Pathologic complete response defined as the absence of tumor cells assessed on the surgical specimen + residual Ductal Carcinoma In Situ (DCIS) in the breast.

SECONDARY OUTCOMES:
Determine predicting factors at the phosphoproteomic signature and its correlation with response to BIBF-1120 | Baseline and end of priming phase.
  1. Determination of phosphoproteomic signatures in tumor biopsy. Patients in arm-2 will undergo a baseline biopsy with the aim of establishing a signature predicting response to docetaxel alone, and by comparison with the signature in the arm-1, extracting the signalling nodes implicated in docetaxel response from those implicated in angiogenic blockade response.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ángel Quintela, M.D.,PhD, Study Director — CNIO; Ramón Colomer, M.D.,PhD, Principal Investigator — CNIO
Locations (3):
- Spain (3):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - MD Anderson Cancer Centre Madrid, Madrid